CLINICAL TRIAL: NCT01774890
Title: ST2, a Novel Biomarker for Cardiac Remodeling in Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Amiram Nir, Head, Adult Congenital Heart Disease Unit, Hadassah Medical Organization
Other Study IDs: 0599-12-HMO
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The remarkable improvement in survival of children with congenital disease has led to a continuously growing number of adults with congenital heart disease in the developed world. Many of these patients had had cardiac surgery at early age, the may live for many years with pressure overload, volume overload, systolic or diastolic dysfunction, cyanosis or any combination of the above. These past and ongoing cardiac insults often result in significant cardiac remodeling. A biomarker for fibrosis and remodeling may have enormous clinical and prognostic value for these patients.

Serum biomarkers are now integrated in many fields in medicine. In cardiology, a number of biomarkers are used. In the last decade, our group has focused on the natriuretic peptides as markers for heart disease in infants and children. This resulted in many studies and more than 25 publications in the medical literature. We believe that the newly discovered cardiac marker, ST2, will emerge as an important addition to cardiac evaluation in the coming years.The aim of this study is to measure ST2 levels in patients with congenital right heart disease and correlate ST2 levels to clinical status, imaging and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age>18 y)
* congenital heart disease

Exclusion Criteria:

* Additional lung diseases, renal disease or inflammatory disease.
* Patients who underwent therapeutic intervention between the MRI and the ST2 - measurements.
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults born with congenital heart disease in stable clinical condition
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
NYHA classification and/or 6 minute walk distance | six months

SECONDARY OUTCOMES:
Hemoglobin level | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizrtion, Jerusalem, Israel